CLINICAL TRIAL: NCT06528015
Title: Efficacy and Safety of Probiotics Combined With Enteric-coated Budesonide Capsules in Patients With Primary IgA Nephropathy: a Prospective, Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Probiotics Combined With Enteric-coated Budesonide Capsules in Patients With Primary IgA Nephropathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gang Xu (Other)
Collaborators: China Primary Health Care Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Gang Xu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TongjiHospitalxugangtjh123
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Glomerulonephritis, IGA; Probiotics; Budesonide
Keywords: enteric-coated budesonide capsules; probiotic; primary IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Experimental participants will receive probiotics combined with enteric-coated budesonide capsules
  Interventions: Drug: probiotics combined with enteric-coated budesonide capsule
- Comparator (Placebo Comparator): Comparator participants will receive probiotics placebo combined with enteric-coated budesonide capsules
  Interventions: Drug: probiotics placebo combined with enteric-coated budesonide capsules

INTERVENTIONS:
Drug: probiotics combined with enteric-coated budesonide capsule — In the 9-month treatment period, the following treatments will be received: probiotics combined with enteric-coated budesonide capsules group: 1 bag/day of probiotics (each bag added active probiotic Lactobacillus casei Zhang ≥100 billion CFU) +16 mg/day oral enteric-coated budesonide capsules.
  After completing the treatment period, participants will enter a 2-week reduction period to reduce the risk of adrenal insufficiency. ① enteric-coated budesonide capsules reduction: 8 mg/day oral enteric-coated budesonide capsules.
  Arms: Experimental
Drug: probiotics placebo combined with enteric-coated budesonide capsules — In the 9-month treatment period, the following treatments will be received: probiotics placebo combined with enteric-coated budesonide capsules group: 1 bag/day of probiotics placebo +16 mg/day oral enteric-coated budesonide capsules.
  After completing the treatment period, participants will enter a 2-week reduction period to reduce the risk of adrenal insufficiency. ① enteric-coated budesonide capsules reduction: 8 mg/day oral enteric-coated budesonide capsules.
  Arms: Comparator

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of probiotics combined with enteric-coated budesonide capsule in patients with IgA nephropathy on the basis of optimized RAS blockade therapy, and to explore the correlation between the efficacy of probiotics combined with enteric-coated budesonide capsule in the treatment of primary IgA nephropathy and intestinal homeostasis.

The main questions it aims to answer are:

Dose probiotics combined with enteric-coated budesonide capsule provide a durable reduction in urine protein creatinine ratio (UPCR) in participants, compared with probiotics placebo combined with enteric-coated budesonide capsule? What medical problems do participants have when taking probiotics combined with enteric-coated budesonide capsule?

Participants will:

Take probiotics combined with enteric-coated budesonide capsules or probiotics placebo combined with enteric-coated budesonide capsules every day for 9.5 month Participate in center site follow-up visits for 13 times Keep a diary of their symptoms and outcomes

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, single-blind, placebo-controlled clinical trial. The study included a screening period (7-15 days), an induction period (at least 3 months), randomization, a treatment period (9 months), a reduction period (2 weeks), a safety follow-up period (2.5 months), and a long-term follow-up period (36 months). Participants who meet the randomization criteria will be randomly assigned (1:1) to receive probiotics combined with enteric-coated budesonide capsules or probiotics placebo combined with enteric-coated budesonide capsules.

Screening period (7-15 days): Participants who sign the informed consent for this study and undergo relevant examinations can enter the induction period if they meet the screening criteria.

Induction period (at least 3 months): Optimized treatment with RAS blockers is performed immediately upon entry the induction period.

Randomization: RAS blockers were used for at least 3 months during the induction period. All inclusion conditions had to be met to qualify for randomization.

Treatment period (9 months): Participants who meet the randomization criteria will be randomly assigned (1:1) to receive probiotics combined with enteric-coated budesonide capsules group or probiotics placebo combined with enteric-coated budesonide capsules. In the 9-month treatment period, the following treatments will be received: ① probiotics combined with enteric-coated budesonide capsules group: 1 bag/day of probiotics (each bag added active probiotic Lactobacillus casei Zhang ≥100 billion CFU) +16 mg/day oral enteric-coated budesonide capsules. ② probiotics placebo combined with enteric-coated budesonide capsules group: 1 bag/day of probiotics placebo +16 mg/day oral enteric-coated budesonide capsules.

The RAS blocker (ACEI or ARB) dosing regimen needs to be stable during treatment period.

Reduction period (2 weeks): After completing the treatment period, participants will enter a 2-week reduction period to reduce the risk of adrenal insufficiency. ① enteric-coated budesonide capsules reduction: 8 mg/day oral enteric-coated budesonide capsules.

The RAS blocker (ACEI or ARB) dosing regimen needs to be stable during reduction period.

Safety follow-up period (2.5 months): After completion of the reduction period, all participants stopped taking the investigational drug, completed the remainder of the safety follow-up period. During this time, the RAS blocker (ACEI or ARB) dosing regimen needs to be stable.

Long-term follow-up period (36 months): Participants who have completed the treatment period, reduction period, and safety follow-up period, as well as those who terminated the study treatment early but did not withdraw from the study, will enter long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age: 18~70 years old;
2. Renal biopsy-confirmed primary IgA nephropathy;
3. 24-h urine protein excretion ≥ 0.75g, or urinary protein creatinine ratio (UPCR) ≥ 0.5g/g;
4. eGFR ≥ 30mL/min/1.73m^2 estimated with the Chronic Kidney Disease Epidemiology Collaboration 2009 formula (CKD-EPI2009);
5. Fertile men and female of childbearing age need to use highly effective contraceptive measures from the time they sign informed consent to the end of the safety follow-up period;
6. Sign the informed consent, understand and agree to comply with the requirements of the study and the trial procedures.

Exclusion Criteria:

1. Secondary form of IgA nephropathy or any non-IgA nephropathy Glomerulonephritis;
2. Specific types of IgA nephropathy (including minor lesions with mesangial IgA deposition, rapidly progressive and crescentic IgA nephropathy, etc.) and other glomerular diseases (such as diabetic nephropathy, etc.);
3. 24-h urine protein excretion >5g;
4. Renal biopsy showed crescent ≥25%;
5. A history of severe gastrointestinal disease (such as active peptic ulcer disease, active gastrointestinal bleeding, gastrointestinal perforation, inflammatory bowel disease, and chronic diarrhea) or a history of gastrointestinal surgery;
6. Complicated with malignant tumors (diagnosed within the past 5 years), cerebral infarction, cerebral hemorrhage, myocardial infarction, arrhythmia, heart failure and other serious primary diseases;
7. The presence of severe chronic or active infections (including but not limited to tuberculosis) that require systemic antimicrobial, antifungal, antiviral, or antiparasitic treatment;
8. A history of cirrhosis;
9. Severe osteoporosis requiring treatment;
10. Received organ transplants;
11. Glaucoma or cataracts who currently require clinical treatment;
12. Diagnosed with uncontrolled mental illness;
13. Participants with poorly controlled type 1 or type 2 diabetes (glycated haemoglobin [HbA1c] >8%;
14. Laboratory tests for abnormal liver function (ALT and/or AST> 2 times the upper normal limit, ALP> 2.5 times the upper normal limit);
15. The blood total cholesterol was seriously abnormal (>12.92mmol/L);
16. Human immunodeficiency virus antibody positive, treponema pallidum antibody positive, hepatitis B surface antigen positive, hepatitis C antibody positive;
17. Currently using a potent inhibitor of cytochrome P4503A4 (CYP3A4) and cannot be discontinued during the study;
18. Known allergy or intolerance to ACEI, ARB, budesonide or any component of the investigational drug formulation;
19. Use of antibiotics, glucocorticoids or other immunosuppressants, foods and medicines containing probiotics/prebiotics within the past 3 months;
20. Pregnant or lactating participants;
21. Also accepting participants from other clinical trials;
22. Participants who have been determined by the researchers to be unable to complete on time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
UPCR | over the 9-month treatment phase
  Mean change from baseline in UPCR over the 9-month treatment phase

SECONDARY OUTCOMES:
UPCR | at 12 months
  Mean change from baseline in UPCR at 12 months
24-h urine protein excretion | at 9 and 12 months
  Mean changes from baseline in 24-h urine protein excretion at 9 and 12 months
UACR | at 9 and 12 months
  Mean changes from baseline in UACR at 9 and 12 months
serum Gd-IgA1 | at 3, 6, 9 and 12 months
  Mean changes from baseline in serum Gd-IgA1 at 3, 6, 9 and 12 months
serum BAFF and APRIL | at 12 months
  Mean changes from baseline in serum BAFF and APRIL at 12 months
eGFR | at 9 and 12 months
  Mean changes from baseline in eGFR at 9 and 12 months
eGFR | 12months，24months，36months after the end of treatment
  Changes from baseline in eGFR at each visit during long-term follow-up
UACR | 12months，24months，36months after the end of treatment
  Changes from baseline in UACR at each visit during long-term follow-up
24-h urine protein excretion | 12months，24months，36months after the end of treatment
  Changes from baseline in 24-h urine protein excretion at each visit during long-term follow-up
renal function (including creatinine, urea, and uric acid) | 12months，24months，36months after the end of treatment
  Changes from baseline in renal function (including creatinine, urea, and uric acid) at each visit during long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GANG XU, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China